CLINICAL TRIAL: NCT05140915
Title: Vaper to Vaper: A Multimodal Mobile Peer Driven Intervention to Support Adolescents in Quitting Vaping
Acronym: V2V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajani Sadasivam, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H00021082; R34DA050992 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2021-12-02 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: E-cigarette Use; Vaping
Keywords: Vaping; Adolescents
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Students in schools randomized to the intervention will receive: (1) peer messages, written by current and former adolescent e-cigarette users and tailored by age and readiness-to-quit; (2) peer coaching, facilitated by texting; and (3) gamification, designed to motivate participation.
  Interventions: Behavioral: Peer Messaging; Behavioral: Peer Coaching via Text; Behavioral: Gamification
- Control (Active Comparator): Students in schools randomized to the control condition will be provided e-cigarette cessation materials by the Research Coordinator at the time of study enrollment.
  Interventions: Other: E-Cigarette Cessation Materials

INTERVENTIONS:
Behavioral: Peer Messaging — Peer messages, written by current and former adolescent e-cigarette users and tailored by age and readiness-to-quit.
  Arms: Intervention
Behavioral: Peer Coaching via Text — Peer coaching, facilitated by texting
  Arms: Intervention
Behavioral: Gamification — Gamification, designed to motivate participation
  Arms: Intervention
Other: E-Cigarette Cessation Materials — E-cigarette cessation materials by the Research Coordinator at the time of study enrollment.
  Arms: Control

SUMMARY:
The dramatic increase in the use of e-cigarettes among U.S. adolescents has been called a national epidemic, with more adolescents now using e-cigarettes than traditional cigarettes. The high amounts of nicotine in e-cigarettes harm adolescents and put them at greater risk of becoming traditional cigarette smokers. The investigators propose to develop Vaper-to-Vaper (V2V), a suite of mobile peer driven tools including peer texting and coaching based on lessons learned in the investigators' prior tobacco intervention work, to engage and help adolescents use strategies to manage cravings and successfully quit.

DETAILED DESCRIPTION:
The FDA and the US Surgeon General call the increasing use of e-cigarettes among U.S. adolescents an epidemic, with e-cigarette use exceeding combustible cigarette use. The high amounts of nicotine in e-cigarettes harm adolescent brain development, impacting learning, memory, and attention. Adolescent e-cigarette users also are at higher risk than non-users of transitioning to traditional cigarettes. While prevention is important, evidence-based interventions to engage and help adolescent e-cigarette users quit are critically needed. Key challenges include adolescents perceiving e-cigarette use to be of low risk resulting in a low intention to quit, and the major influence of peers in e-cigarette use. Given there currently are no evidence-based cessation interventions to assist adolescent e-cigarette users in quitting, as suggested by the American Academy of Pediatrics and FDA, the investigators propose to develop Vaper-to-Vaper (V2V), a multi-modal mobile peer driven intervention, based on lessons learned in our prior tobacco intervention work. Peer-driven interventions have been found to successfully improve smoking outcomes in adolescents, and the investigators have had success in developing peer-driven interventions for low motivated adult smokers. The Investigators therefore will adapt these approaches for adolescent e-cigarette users. V2V's goal will be to engage, educate, motivate, and facilitate the adolescent in using strategies to manage cravings and successfully quit. The V2V components will include: Peer Messaging (tailored messages pushed via texting), Peer Coaching (asynchronous communications with trained coaches via texting), and Gamification (using game design to motivate participation). Adapting these tools to the unique needs of adolescent e-cigarette users will further extend these tools into novel directions. For Aim 1 the investigators will convene a peer advisory panel of 20 adolescent e-cigarette users to participate in a qualitative assessment and further development of V2V components. In Aim 2 the investigators will evaluate the feasibility of the research protocols and the feasibility and acceptability of the V2V intervention in a pilot feasibility study with eighty adolescent e-cigarette users from 4 high schools (schools randomized to either V2V intervention or control) recruited and followed for 6 months. The investigators hypothesize being able to recruit 80 adolescents (20/school, 40 per study condition) and that >85% will be retained in each study condition at 6-month follow-up (Aim 2A). For Aim 2b the investigators will monitor V2V engagement (e.g., number of V2V texting quizzes completed, peer coaching interactions, peer videos viewed) and assess acceptability of and satisfaction with the program. For Aim 2C the investigators hypothesize that the intervention will be associated with greater cotinine-validated 7-day point prevalence vaping abstinence rates, lower time to first quit attempt, and less amount of e-cigarette use compared to control at 6-month follow-up. This Stage I project, adapting an existing intervention and feasibility/pilot testing, will provide the necessary materials and information to proceed to a subsequent large-scale Stage III R01 trial to test the efficacy of the V2V intervention in supporting adolescent e-cigarette users in quitting.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in grade 9-12 at participating high school
* Current e-cigarette user, as defined as a response greater than "0 days" to the question: "During the past 7 days, on how many days did you use e-cigarettes?" This eligibility criterion is modeled on a question in the 2018 National Youth Tobacco Survey (NYTS), a survey of U.S. middle and high school students which used a 30-day timeframe.
* Have a smartphone.
* English- or Spanish-speaking

Exclusion Criteria: Unable or unwilling to provide informed assent or consent (in the case of those aged 18 years or older).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajani Sadasivam, PhD, Principal Investigator — University of Massachusetts Chan Medical School; Lori Pbert, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The final dataset will be available within 12 months of the end of the funded grant period. Due to the nature of our research, we will be collecting identifying information (i.e. names, phone numbers). We will strip the final dataset of identifiers prior to release for sharing. Even though the final dataset will be striped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of study participants with unusual characteristics. Thus, we will make the data and associated documentation available to qualified academic investigators for non-commercial research under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Pbert L, Dube CE, Nagawa CS, Simone DP, Wijesundara JG, Sadasivam RS. Vaping cessation support recommendations from adolescents who vape: a qualitative study. BMC Public Health. 2024 Jun 17;24(1):1615. doi: 10.1186/s12889-024-19036-1. PMID 38886719
- [Derived] Pbert L, Dube CE, Nagawa CS, Simone DP, Wijesundara J, Sadasivam R. Vaping Cessation Support Recommendations from Adolescents Who Vape: A Qualitative Study. Res Sq [Preprint]. 2024 Mar 20:rs.3.rs-4077848. doi: 10.21203/rs.3.rs-4077848/v1. PMID 38562810

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Groups:
- Intervention: Schools were randomized to either the intervention or control condition. Students in schools randomized to the intervention received: (1) peer messages, written by current and former adolescent e-cigarette users and tailored by age and readiness-to-quit; (2) peer coaching, facilitated by texting; and (3) gamification, designed to motivate participation.
- Control: Schools were randomized to either the intervention or control condition. Students in schools randomized to the control condition were provided written e-cigarette cessation materials by the Research Coordinator at the time of study enrollment.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 39; 3 Schools | 32; 2 Schools
Completed | 37; 3 Schools | 31; 2 Schools
Not Completed | 2; 0 Schools | 1; 0 Schools
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Students in school randomized to the intervention will receive: (1) peer messages, written by current and former adolescent e-cigarette users and tailored by age and readiness-to-quit; (2) peer coaching, facilitated by texting; and (3) gamification, designed to motivate participation.
  Peer Messaging: Peer messages, written by current and former adolescent e-cigarette users and tailored by age and readiness-to-quit.
  Peer Coaching via Text: Peer coaching, facilitated by texting
  Gamification: Gamification, designed to motivate participation
- Control: Students in schools randomized to the control condition will be provided written e-cigarette cessation materials by the Research Coordinator at the time of study enrollment. The written materials will consist of two pamphlets from Journeyworks, selected based on: (1) their clear and attractive layout designed for a low-literacy audience, and (2) their providing both information re: e-cigarette use with a strong message about nicotine and nicotine addiction, E-Cigarettes: 8 Things Everyone Should Know, and support in quitting, How to Quit Vaping.
  E-Cigarette Cessation Materials: Written e-cigarette cessation materials by the Research Coordinator at the time of study enrollment. The written materials will consist of two pamphlets from Journeyworks, selected based on: (1) their clear and attractive layout designed for a low-literacy audience, and (2) their providing both information re: e-cigarette use with a strong message about nicotine and nicotine addiction, E-Cigarettes: 8 Things Everyone Should Know, and support in quitting, How to Quit Vaping.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 39 | 32 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 24 | 47
  Between 18 and 65 years | 16 | 8 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.3 (1.2) | 16.8 (1.0) | 17.07 (1.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Non-Binary | 1 | 0 | 1
  Transgender | 1 | 0 | 1
  Male | 17 | 16 | 33
  Female | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 15 | 20
  Not Hispanic or Latino | 29 | 16 | 45
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 29 | 18 | 47
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 32 | 71
Grade [Count of Participants; unit: Participants]
  9th | 6 | 3 | 9
  10th | 6 | 17 | 23
  11th | 12 | 8 | 20
  12th | 15 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Participant Recruitment and Retention
Description: Investigators will assess the number of those screened, eligible, and consented who remain active in the program at 3 months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 39 | 32
Participants | 37 | 31

2. Secondary Outcome: Acceptability of and Satisfaction With the Intervention
Description: Investigators will access the acceptability of and satisfaction with the intervention, as measured by Client Satisfaction Questionnaire (CSQ-8).The overall CSQ-8 score is calculated by summing the respondent's rating (item rating) score for each scale item. Scores therefore range from 8 to 32, with higher values indicating higher satisfaction. Similarly, investigators will look for association between summary score and cessation.
Time Frame: 3 months
Population: The data for this outcome measure were based on participant self-report. As participants were not required to answer all survey questions, the number of participants analyzed reflects only those who responded to the specific questions related to this outcome on the surveys.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 32 | 20
scores on a scale | 25.34 (4.65) | 24.95 (4.64)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .77, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Abstinence From Vaping as Measured by Saliva Samples [Cotinine-validated 7-day Point Prevalence]
Description: Cotinine-validated 7-day point prevalence abstinence, as measured by saliva samples collected from all; analyzed for those reporting 7-day abstinence; cut-off 11.4 ng/ml, cotinine-imputed abstinence when cotinine is missing.
Time Frame: 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 32
Participants | 5 | 5

4. Secondary Outcome: Number of Peer Coaching Interactions
Description: Investigators will assess the system use (for V2V intervention only), as measured by the number of peer coaching interactions completed.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Number of interactions
Arm/Group | Intervention
Number analyzed (Participants) | 37
Number of interactions | 5.05 (4.59)

5. Secondary Outcome: Number of Peer Videos Viewed
Description: Investigators will assess the system use (for V2V intervention only), as measured by the self-reported frequency of viewing peer videos.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 37
Participants
  Never | 12
  Very Rarely (Once) | 10
  Rarely (1-2 days/week) | 6
  Occasionally (3-4 days/week) | 5
  Frequently (5 days/week) | 2
  Very Frequently | 0
  Prefer not to answer | 2

6. Secondary Outcome: Number of Games Engaged In
Description: Investigators will assess the system use (for V2V intervention only), as measured by the self-reported frequency of reading gamification texts.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 37
Participants
  Always | 6
  Usually | 6
  About half the time | 6
  Rarely | 10
  Never | 8
  Prefer not to answer | 1

7. Secondary Outcome: Change in Self-Efficacy Score
Description: Assessment of change in self-efficacy, as measured by the Self-efficacy Questionnaire (SEQ-12). The SEQ-12 (Self-Efficacy) Score is the mean of 12 items coded 1 (Not at all confident) to 5 (Extremely Confident). The score can range from 1-5, with higher scores indicating better confidence to refrain from vaping.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 31
scores on a scale | -.19 (.20) | .15 (.22)

8. Secondary Outcome: Number of Participants With With Change in Stage of Change
Description: Investigators will also assess the change in stage of change, as measured by Prochaska's Stages of Change model. The stages of change are: Precontemplation, Contemplation, Preparation/Determination, Action/Willpower, Maintenance, and Relapse. Participants will self-report their stage of change at 0 and 3 months.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 30
Participants
  Worse | 5 | 6
  Same | 15 | 17
  Better | 14 | 7

9. Secondary Outcome: Change in Severity of Nicotine Addiction
Description: Investigators will assess the change in the severity of nicotine addiction, as measured by the Hooked on Nicotine Checklist. The Hooked on Nicotine Checklist Score is the sum of 10 items coded 0 (Not endorsed) or 1 (Endorsed). The possible range is 0-10, with higher scores indicating a higher level of addiction.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 31
scores on a scale | -.37 (.79) | -1.19 (.87)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 3 months (participants' duration in the study).
Description: For this study, the standard Adverse Event and Serious Adverse Event definitions were used.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/32
Other Adverse Events (participants affected / at risk) | 0/39 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05140915/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT05140915/ICF_001.pdf